CLINICAL TRIAL: NCT01112709
Title: Maintaining Resistance Training in Older Prediabetic Adults: Theoretical Approach
Brief Title: Maintaining Resistance Training in Older Prediabetic Adults
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Virginia Polytechnic Institute and State University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Brenda Davy, Associate Professor, Virginia Polytechnic Institute and State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 1R01DK082383-01A1 (NIH); R01DK082383 (NIH)
Record Dates: First submitted 2010-04-22; First posted 2010-04-28 (Estimated); Last update posted 2014-03-20 (Estimated); Status verified 2014-03

CONDITIONS: Diabetes; Prediabetes
Keywords: Diabetes; Prediabetes; Resistance training; behavior; behavioral change theory
MeSH Terms: conditions — Diabetes Mellitus; Prediabetic State; Behavior

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- SCT (Experimental): This arm is a long-term, Social Cognitive Theory (SCT)-based intervention, emphasizing self-regulation and other SCT strategies to optimize training, with faded contact.
  Interventions: Behavioral: SCT-based Resistance Training exercise program
- Control (Active Comparator): This arm will be the "control" condition; a Standard intervention with minimal contact.
  Interventions: Other: Standard Intervention with minimal contact

INTERVENTIONS:
Behavioral: SCT-based Resistance Training exercise program — Two supervised RT sessions per week for the first 3 months, then a self-monitored RT phase for the remainder of the study, with primarily Internet-based contact.
  Arms: SCT
Other: Standard Intervention with minimal contact — This is the control condition for comparison; the approach will be identical to the experimental condition, but without the theoretical components (skills to increase self efficacy for RT, self regulation for RT). Contact with the study staff will be reduced from that received by the experimental group.
  Arms: Control

SUMMARY:
The aim of this Phase II Clinical Trial is to demonstrate the efficacy of social cognitive theory (SCT) based intervention for initiating, and most importantly, maintaining resistance training in older adults with pre-diabetes (i.e., impaired glucose tolerance or impaired fasting glucose) to improve blood glucose regulation.

DETAILED DESCRIPTION:
The aim of this Phase II Clinical Trial is to demonstrate the efficacy of social cognitive theory (SCT) based intervention for initiating, and most importantly, maintaining resistance training in older adults with pre-diabetes (i.e., impaired glucose tolerance or impaired fasting glucose) to improve glucose homeostasis. The overall aim is consistent with NIDDK's Behavioral/Prevention Research Program's focus on individual, family, and community-based strategies for prevention of diabetes and its complications. Resistance training is particularly applicable to older, pre-diabetic adults given the loss of lean body mass and worsening of glucose tolerance with aging. The proposed research program evaluates a 15-month SCT based intervention for maintenance of resistance training with older adults. Men and women 50-69 (N=180) with pre-diabetes, defined as exhibiting either impaired glucose tolerance (IGT; 2-h glucose 140-199 mg/dl) or impaired fasting glucose (IFG; 100-125 mg/dl), will first follow the same standard, supervised 3-month initiation period with resistance training. All people completing the Initial Phase will be randomly assigned to 1 of 2 maintenance conditions: 1. a long-term SCT based, ASPIRE intervention, emphasizing self-regulation and other SCT strategies to optimize training, with faded contact; 2. a Standard intervention with minimal contact. The primary outcome measures are indices of pre-diabetes (glucose tolerance and fasting glucose concentration) and strength. Secondary measures include adherence; ß-cell responsivity, insulin sensitivity, and disposition index, as determined by the oral glucose and C-peptide minimal model; fat free mass, other indicators of health and metabolic fitness, and SCT measures. Assessments will occur at baseline, at the end of the Initiation Phase (3 months), at the end of the different interventions (9 months) and 6 months after all contact has ended (15 months from baseline). It is hypothesized that SCT based resistance training with faded contact will produce better outcomes than the Standard-based resistance training at 9 month and 15 month assessments. It also is hypothesized that improvements in glucose homeostasis and in strength from resistance training will be mediated by adherence, self-efficacy, and use of self-regulation strategies. Resistance training has become an important component in the treatment and prevention of diseases and disabilities, and especially so for Type 2 diabetes. Critical to public health and a focus of NIDDK are theory-based interventions that enable, effective long-term resistance training with minimal supervision after an initiation phase and where improvements in adherence and outcomes are facilitated by theoretical constructs.

ELIGIBILITY:
Inclusion Criteria:

* prediabetes,
* overweight or obese,
* aged 50-69 years,
* otherwise good health,
* physician clearance for exercising,
* sedentary (< 150 min/wk of moderate intensity physical activity).

Exclusion Criteria:

* diagnosed with diabetes or other conditions that would preclude an individual from safely resistance training (eg, heart disease),
* currently engaging in RT (for > 1 year),
* smokers,
* uncontrolled hypertension,
* retinopathy,
* recent cataract surgery,
* recent head trauma.

Ages: 50 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Actual)
Dates: Start 2011-01; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Markers of prediabetes | 15 months
  glucose tolerance and fasting glucose concentration
Muscular Strength | 15 months
  3 RM (repetition maximum - the maximum amount of weight that can be lifted three times)

SECONDARY OUTCOMES:
Insulin secretion and action | 15 Months
Adherence to the resistance training program session schedule (twice/week sessions) | 15 Months
Social Cognitive Theory Measures (includes self-efficacy, self-regulation, outcome expectancies, and affect; related to resistance training) | 15 Months
Body Composition | 15 Months

CONTACTS AND LOCATIONS:
Overall Officials: Brenda M Davy, PhD, RD, Principal Investigator — Virginia Polytechnic Institute and State University; Richard A Winett, PhD, Principal Investigator — Virginia Polytechnic Institute and State University
Locations (2):
- United States (2):
  - Virginia Tech, Blacksburg, Virginia
  - VT Riverside, Roanoke, Virginia

REFERENCES:
- [Derived] Davy BM, Winett RA, Savla J, Marinik EL, Baugh ME, Flack KD, Halliday TM, Kelleher SA, Winett SG, Williams DM, Boshra S. Resist diabetes: A randomized clinical trial for resistance training maintenance in adults with prediabetes. PLoS One. 2017 Feb 23;12(2):e0172610. doi: 10.1371/journal.pone.0172610. eCollection 2017. PMID 28231265
- [Derived] Eikenberg JD, Savla J, Marinik EL, Davy KP, Pownall J, Baugh ME, Flack KD, Boshra S, Winett RA, Davy BM. Prediabetes Phenotype Influences Improvements in Glucose Homeostasis with Resistance Training. PLoS One. 2016 Feb 3;11(2):e0148009. doi: 10.1371/journal.pone.0148009. eCollection 2016. PMID 26840904
- [Derived] Halliday TM, Davy BM, Clark AG, Baugh ME, Hedrick VE, Marinik EL, Flack KD, Savla J, Winett S, Winett RA. Dietary intake modification in response to a participation in a resistance training program for sedentary older adults with prediabetes: findings from the Resist Diabetes study. Eat Behav. 2014 Aug;15(3):379-82. doi: 10.1016/j.eatbeh.2014.04.004. Epub 2014 May 10. PMID 25064285